CLINICAL TRIAL: NCT01541332
Title: A Phase 1/2 Study of Pomalidomide, Dexamethasone and Pegylated Liposomal Doxorubicin for Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Pomalidomide, Dexamethasone and Pegylated Liposomal Doxorubicin for Relapsed/Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oncotherapeutics (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PO-MM-PI-0049; PDD-2011 (Other: Oncotherapeutics)
Record Dates: First submitted 2012-02-20; First posted 2012-02-29 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Multiple Myeloma
Keywords: relapsed refractory; multiple myeloma; pomalidomide; Doxil; dexamethasone; Oncotherapeutics
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; liposomal doxorubicin; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pomalidomide + PLD + Dexamethasone (Experimental): Pomalidomide + Pegylated Liposomal Doxorubicin + Dexamethasone in an open label, dose escalation study
  Interventions: Drug: Pomalidomide; Drug: Pegylated Liposomal Doxorubicin (PLD); Drug: Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide — Pomalidomide administered to 3 cohorts of subjects at escalating doses of 2 (cohort 1), 3 (cohort 2) and 4 mg/dose (cohort 3) per orem (PO). Doses are to be administered once-a-day, for the first 21 days, as part of a 28-day treatment cycle, followed by a 7-day rest period.
  Other Names: CC-4047
Drug: Pegylated Liposomal Doxorubicin (PLD) — Dexamethasone will be given at a dose of 40 mg/dose IV. Doses are to be administered on days 1, 4, 8, and 11 of the 28-day cycle.
  PLD will be given at a dose of 5.0 mg/m2 as a 60 minute IV infusion on Day 1 of Cycle 1 and subsequent doses may be administered over 30 to 60 minutes on Days 4, 8 and 11 of Cycle 1 and on Days 1, 4, 8, and 11 of each subsequent cycle.
  Other Names: Doxil
Drug: Dexamethasone — Dexamethasone will be given at a dose of 40 mg/dose IV. Doses are to be administered on days 1, 4, 8, and 11 of the 28-day cycle.
  Other Names: Decadron

SUMMARY:
The purpose of this clinical research study is to evaluate the safety and effectiveness (good and bad effects) of a combination of three different drugs, pomalidomide, pegylated liposomal doxorubicin, and dexamethasone when used to treat relapsed (the disease came back) or refractory (the disease did not respond to past treatment) multiple myeloma. Different dosages (amount of study drug) of pomalidomide are first being tested to determine if there are any side effects or risks associated with combining this study drug with the other two listed. Once the optimal dose is decided on, the study will change its focus to determining the effectiveness of the study drug in this combination.

DETAILED DESCRIPTION:
This is a phase 1/2, multicenter, open label and nonrandomized study to evaluate the efficacy and safety of pomalidomide at daily dosages of 2, 3 or 4 mg in combination with intravenous (IV) dexamethasone at 40 mg/dose and Pegylated Liposomal Doxorubicin (PLD) at 5 mg/m2/dose for subjects with relapsed/refractory multiple myeloma (MM). The study consists of a screening period, followed by up to eight 28 day open label treatment cycles, a final assessment to occur 28 days after the end of the last treatment, and a follow-up period.

Subjects eligible for this study will receive treatment with study drug for a maximum of eight 28 day treatment cycles. Subjects are to be treated to a maximum response plus 2 additional cycles (no more than 8 cycles will be allowed) or complete 8 cycles of therapy without disease progression.

Pomalidomide, dexamethasone and PLD will be administered on the appropriate cycle days as shown below.

Cohort 1 Pomalidomide* - 2 mg, Dexamethasone** - 40 mg, PLD** - 5 mg/m2

Cohort 2 Pomalidomide* - 3 mg, Dexamethasone** - 40 mg, PLD** - 5 mg/m2

Cohort 3 Pomalidomide* - 4 mg, Dexamethasone** - 40 mg, PLD** - 5 mg/m2

* PO Days 1-21

** IV Days 1, 4, 8 and 11

In all cohorts, if an unacceptable dose limiting toxicities (DLT) is not seen in any of the 3 subjects during the first cycle of any dose level, dose escalation will continue. All subjects in a cohort must complete a minimum of 28 days or a full cycle, whichever is longer, without a DLT before enrollment to the next cohort can begin. If a DLT is identified in 1 subject at any dose level during the first treatment cycle, an additional 3 subjects will be recruited to this dose level. A maximum of 6 subjects may be enrolled in each cohort. If an unacceptable DLT is observed in 2 subjects at any dose level, no further subjects will be recruited to this dose level. The maximum tolerated dose (MTD) will be declared as the highest dose level at which fewer than 33% of subjects experienced an unacceptable DLT. If pomalidomide at 4 mg is reached and fewer than 33% of subjects experience an unacceptable DLT, 4 mg will be accepted as the putative MTD. Once the MTD is established, further enrollment will continue to expand that dose cohort until the total sample size of 40 subjects is reached for the entire study. During the phase 2 portion of this study, subjects enrolled will have relapsed/refractory MM resistant to lenalidomide as demonstrated by progressive disease while on lenalidomide or that has relapsed within 8 weeks of the last dose of lenalidomide.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MM based on standard criteria (Durie 1986)
* Currently has MM with measurable disease, defined as:

  * a monoclonal immunoglobulin spike on serum electrophoresis of at least 0.5 g/dL and/or
  * urine monoclonal protein levels of at least 200 mg/24 hours
  * for patients without measurable serum and urine M-protein levels, an abnormal free light chain ratio (normal value: 0.26 - 1.65)
* Currently has progressive MM that has relapsed or is refractory, defined as:

  * For the phase 1: Relapsed following stabilization or a response to at least one anti-myeloma regimen or refractory defined as progressed while receiving an anti-myeloma treatment
  * For the phase 2: Refractory to lenalidomide as demonstrated by progressive disease while on lenalidomide or that relapsed within 8 weeks of the last dose of lenalidomide either as a single agent or in combination.
  * Prior treatment with four days or less of a total of 400 mg of prednisone (or an equivalent potency of another steroid) for MM will not be considered a regimen
* Able to adhere to the study visit schedule and other protocol requirements
* ECOG performance status of 2 or greater at study entry
* Life-expectancy of greater than 3 months
* Lab tests within study ranges at study entry:

  * Absolute neutrophil count > 1.5 x 109/L
  * Platelet count > 75 x 109/L
  * Hemoglobin > 8 g/dL
  * Calculated or measured creatinine clearance > 30 mL/minute
  * Total bilirubin < 1.5 x upper limit of normal (ULN)
  * AST (SGOT) and ALT (SGPT) < 2 x ULN
  * Serum potassium within the normal range
* Females of childbearing potential must have a negative serum or urine pregnancy test.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (subjects intolerant to ASA may use warfarin or low molecular weight heparin)

Exclusion Criteria:

* POEMS syndrome
* Plasma cell leukemia
* Primary amyloidosis
* Non-hematologic malignancy within the past 5 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
* Impaired cardiac function or clinically significant cardiac diseases
* Severe hypercalcemia
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the ICF
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Undergone major surgery within 28 days prior enrollment or has not recovered from side effects of such therapy (Kyphoplasty is not considered to be a major surgery; however, the investigator is to discuss enrollment of a subject with a recent history of kyphoplasty with the medical monitor)
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide)
* Received the following prior therapy:

  * Pomalidomide
  * Chemotherapy within 3 weeks of study drugs (6 wks for nitrosoureas)
  * Corticosteroids (>10 mg/day prednisone or equivalent) within 3 weeks of study drugs
  * Immunotherapy or antibody therapy as well as thalidomide, lenalidomide, arsenic trioxide or bortezomib within 21 days before study drugs
  * Extensive radiation therapy within 28 days before study drugs. Receipt of localized radiation therapy does not preclude enrollment.
  * Use of any other experimental drug or therapy within 28 days of study drugs
* Known hypersensitivity to compounds of similar chemical or biological composition to thalidomide, lenalidomide or doxorubicin.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Concurrent use of other anti-cancer agents or treatments
* Known positivity for human immunodeficiency virus (HIV) or hepatitis B or C; baseline testing for HIV and hepatitis B or C is not required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
MTD of Pomalidomide | 12 months
  Phase 1: To establish the MTD of pomalidomide in combination with dexamethasone and pegylated liposomal doxorubicin
Overall Response Rate | 24 months
  Phase 2: To determine efficacy as evidenced by the best overall response rate (CR + VGPR + PR + MR) following treatment with pomalidomide, dexamethasone and pegylated liposomal doxorubicin

SECONDARY OUTCOMES:
Number of Patients with Adverse Events | 24 months
  Phase 2: To establish the number of patients with adverse events when using the combination of pomalidomide, dexamethasone and pegylated liposomal doxorubicin
Time to Progression | 24 Months
  Phase 2: Defined as the time from initiation of therapy to progressive disease
Progression-free Survival | 24 Months
  Phase 2: Defined as the time from initiation of therapy to progressive disease or death from any cause, which ever occurs first
Time to First Response | 24 Months
  Phase 2: Defined as the time from the initiation of therapy to the first evidence of a confirmed response (CR, VGPR, PR or MR)
Duration of Response | 24 Months
  Phase 2: Defined as the time from first response to progressive disease
Overall Survival | 24 Months
  Phase 2: Defined as the time from initiation of therapy to death from any cause or last follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: James R Berenson, MD, Principal Investigator — Oncotherapeutics
Locations (8):
- United States (8):
  - Roy and Patricia Disney Family Cancer Center, Burbank, California
  - California Cancer Associates for Research and Excellence, Encinitas, California
  - Hematology Oncology Medical Group, Fresno, California
  - Pacific Cancer Care, Salinas, California
  - Cancer Center of Santa Barbara, Santa Barbara, California
  - Mission Hope Cancer Center, Santa Maria, California
  - James R Berenson, MD, Inc., West Hollywood, California
  - Illinois Cancer Specialists, Niles, Illinois